CLINICAL TRIAL: NCT03452449
Title: Accelerometry-based Physical Activity, Disability and Quality of Life Before and After Lumbar Spine Surgery: a Prospective Study
Brief Title: Physical Activity, Disability and Quality of Life Before and After Lumbar Spine Surgery
Acronym: PA-LSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00672
Record Dates: First submitted 2018-02-26; First posted 2018-03-02 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Lumbar Spine Degeneration; Physical Activity; Quality of Life; Disability Physical; Pain
Keywords: activity monitor; questionnaire; Oswestry Disability Index
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lumbar spine surgery: Patients undergoing planned lumbar spine surgery
  Interventions: Procedure: planned lumbar spine surgery

INTERVENTIONS:
Procedure: planned lumbar spine surgery — planned lumbar spine surgery including decompression, discectomy, foraminotomy, laminectomy

SUMMARY:
To date it is unknown how physical activity levels in adults is limited before and after lumbar spine surgery and if physical activity level is associated with disability and limitations of quality of life. The main objective is to compare physical activity preoperatively and 6 and 12 weeks postoperatively in patients undergoing lumbar spine surgery with norm data. In addition, the investigators will study the association of changes in physical activity, disability and quality of live.

DETAILED DESCRIPTION:
Patients scheduled for planned lumbar spine surgery will be contacted to participate in this study. All outcomes will be assessed within 1 week preoperatively and at 6 and 12 weeks postoperatively. Changes in outcome scores will be detected using analysis of variance. Association of changes in physical activity and changes in secondary outcomes will be detected using stepwise linear regression models.

ELIGIBILITY:
Inclusion Criteria:

* primary lumbar spine surgery
* single or multi level surgery on segments L2 to S1 (e.g. discectomy, decompression, laminectomy, foraminotomy)
* German speaking

Exclusion Criteria:

* stabilisation or fusion surgery or surgery above L2
* previous lumbar spine surgery
* indication: scoliosis, fracture, trauma, infection, tumor
* limited walking ability due to other conditions
* psychiatric conditions or dementia

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients undergoing planned lumbar spine surgery
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Physical activity | up to 12 weeks
  measured using ActiGraph (accelerometer based activity monitor) as step counts, physical activity intensity during 7-day data capture period

SECONDARY OUTCOMES:
Disability | up to 12 weeks
  measured using Oswestry Disability Index (questionnaire) (best score: 0 - no disability, worst score: 100)
Quality of life assessed by questionnaire | up to 12 weeks
  measured using Short Form (SF)-36 (questionnaire) (worst score: 0; best score: 100 - highest quality of life)
Pain assessed by questionnaire | up to 12 weeks
  measured using 10 cm visual analogue scale (VAS) lower back, legs (best score: 0 - no pain; worst score: 100)

CONTACTS AND LOCATIONS:
Overall Officials: Corina Nüesch, PhD, Study Chair — University Hospital, Basel, Switzerland
Locations (2):
- Switzerland (2):
  - Clinic for Orthopaedics and Traumatology, University Hospital basel, Basel, Canton of Basel-City
  - Bethesda Spital AG, Basel

IPD SHARING:
Plan to Share IPD: No